CLINICAL TRIAL: NCT00620672
Title: To Compare Measures of Central Nervous System Maturity of Visual Acuity, Language, Mental and Motor Skill Development in Term Infants Following Maternal Supplementation Wit the n-3 Fatty Acid Docosahexaenoic Acid (DHA) During Gestation.
Brief Title: N-3 Fatty Acid Requirements for Human Development
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H03-70242; CW03-0084
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy
Keywords: n-3 supplementation during pregnancy; DHA and pregnancy, infant development; n-3 status and gestation; DHA and visual acuity and cognition during infancy
MeSH Terms: interventions — Fatty Acids, Omega-3; Plant Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): The dietary supplement is 400 mg/day of the omega 3 fatty acid docosahexaenoic acid . The docosahexaenoic acid is provided in triglycerides from Martek Biosciences, Maryland. The supplement is a blend of soybean and canola oil, blended to resemble the usual fat composition of the diet. Both the supplement and placebo provide a total of about 10 calories per day to the diet.
  Interventions: Dietary Supplement: omega 3 fatty acids
- 2 (Other): Dietary supplement is vegetable oil, the placebo.
  Interventions: Dietary Supplement: vegetable oil

INTERVENTIONS:
Dietary Supplement: omega 3 fatty acids — The supplements are taken orally with a meal, each day. The amount of the omega 3 fatty acid docosahexaenoic acid is 400 mg/day; taken in two 500 mg capsules each providing 200 mg docosahexaenoic acid. The placebo is two 500 mg capsules soybean/canola oil. Both the supplement and placebo are a total of 1 gm/day (2x500 mg) and about 10 calories per day.
  Arms: 1
Dietary Supplement: vegetable oil — The supplement is a dietary supplement of vegetable oil as a placebo
  Arms: 2

SUMMARY:
Polyunsaturated fatty acids known as n-3 fatty acids are essential dietary nutrients for humans, and are known to be important to reducing the risk of certain diseases, particularly those related to neural system, cardiovascular system and immune system. Among the different n-3 fatty acids, docosahexaenoic acid (DHA) is present in particularly high amounts in the brain and retina, and is accumulated in large amounts in these organs during the last trimester of fetal development and first few months after birth. The n-3 fatty acids are present in the diet as linolenic acid which is found in vegetable and seed oils, and as DHA which is only found in animal tissue fats, with fatty fish being the richest dietary source. Humans are able to convert linolenic acid to DHA, but the conversion is believed to be slow in human and possibly inadequate to support the needs for DHA for the developing brain. Information from our work and those of others has suggested that DHA is important during pregnancy, however specific evidence is lacking to show that the DHA status of pregnant women in low, or that improvement in the DHA status of Canadian women during pregnancy will have benefit to early infant an child development. There is no evidence that infants of vegans and vegetarians, or women who do not eat DHA are at risk for developmental delays. The purpose of this study is to investigate whether a dietary supplement of DHA during pregnancy has any effect on infant birth weight, or indices of infant growth, visual, mental and motor skill development.

DETAILED DESCRIPTION:
This is a randomized, blinded prospective study with 2 groups: placebo and group supplemented with DHA. Women are randomized at 16 weeks gestation without knowledge of their dietary fatty acid intake. Only healthy women expecting to deliver a single infant with no known or anticipated maternal or fetal complications are enrolled. Maternal venous blood is collected at 16 and 36 weeks of gestation and used to assess the maternal DHA status and effect of DHA supplementation. Dietary information is collected at 16 and 36 weeks of gestation to determine usual fatty acid intakes. Following delivery, fetal cord blood is collected to assess transfer of DHA from mother to fetus. Breast milk samples are collected from all breast feeding mothers at 1 and 2 months postpartum. The mother -infant pairs are followed for 18 months. Measures include visual acuity, language, motor and mental development, and growth and dietary intakes.

ELIGIBILITY:
Inclusion Criteria:

* 12-16 weeks gestation
* Low risk pregnancy
* Expected to deliver single full term
* No maternal metabolic or infectious disease
* No known fetal complications.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2004-05; Primary Completion 2011-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Primary outcome is measuring of infant CNS maturity to 18 months of age | 18 months
  Primary outcome is measuring of infant CNS maturity to 18 months of age

SECONDARY OUTCOMES:
Length of gestation and infant birth weight, infant growth (weight, length and head circumference) at 1,2 6,9,12,14,and 18 months Language development at 14 and 16 months | 72 months
  * Length of gestation and infant birth weight, infant growth (weight, length and head circumference) at 1,2 6,9,12,14,and 18 months
  * Diet, blood an dbreast milk fatty acids

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M. Innis, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Mulder KA, King DJ, Innis SM. Omega-3 fatty acid deficiency in infants before birth identified using a randomized trial of maternal DHA supplementation in pregnancy. PLoS One. 2014 Jan 10;9(1):e83764. doi: 10.1371/journal.pone.0083764. eCollection 2014. PMID 24427279
- [Derived] Friesen RW, Innis SM. Linoleic acid is associated with lower long-chain n-6 and n-3 fatty acids in red blood cell lipids of Canadian pregnant women. Am J Clin Nutr. 2010 Jan;91(1):23-31. doi: 10.3945/ajcn.2009.28206. Epub 2009 Nov 18. PMID 19923368
- [Derived] Friesen RW, Innis SM. Dietary arachidonic acid to EPA and DHA balance is increased among Canadian pregnant women with low fish intake. J Nutr. 2009 Dec;139(12):2344-50. doi: 10.3945/jn.109.112565. Epub 2009 Oct 28. PMID 19864401
- [Derived] van Dijk CE, Innis SM. Growth-curve standards and the assessment of early excess weight gain in infancy. Pediatrics. 2009 Jan;123(1):102-8. doi: 10.1542/peds.2007-3382. PMID 19117867